CLINICAL TRIAL: NCT05078307
Title: Evaluation of a Hysteroscopic Method With Vaporization in the Hysteroscopic Treatment of Submucosal Uterine Fibroids
Acronym: VAPOHYSTERO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-09; IDRCB (Other: 2021-A01040-41)
Record Dates: First submitted 2021-09-15; First posted 2021-10-14 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Uterine Fibroids
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OHR System (Active Comparator): Use of the OHR system to perform an operative hysteroscopy by resection of the fibroid.
  Interventions: Procedure: OHR VS OHV
- OHV System (Experimental): Use of the OHV system to perform an operative hysteroscopy by vaporization of the fibroid.
  Interventions: Procedure: OHR VS OHV

INTERVENTIONS:
Procedure: OHR VS OHV — Control group : use of the OHR system to perform an Operative Hysteroscopy by Resection of the fibroid.
  Experimental group : use of the OHV system to perform an Operative Hysteroscopy by Vaporization of the fibroid.

SUMMARY:
Operative hysteroscopy (OH) is an endoscopic technique for the treatment of benign intrauterine lesions and in particular uterine fibroids. The limit of this technique is the duration of the operation which is correlated with the operative risks. Thus, when there is a large fibroid or several fibroids, this technique can sometimes not be used or require several sessions. Today there is a new technique of HO that theoretically allows a gain in operative time. There are few comparative studies showing a clinically interesting gain in operating time. The aim of this study is to compare the operative time between the classical HO technique by resection and the vaporization technique.

This is a randomized, single-center study. The study population corresponded to women aged over 18 years requiring operative hysteroscopy for fibroids. After obtaining informed consent, patients will be randomized into two groups: a vaporization hysteroscopy group and a resection hysteroscopy group. The primary endpoint will be operative time. The secondary endpoints will be intraoperative characteristics and complications (amount of distension fluid used, cervical injury, uterine perforation), immediate postoperative data (pain) and medium-term data (postoperative synechiae). The starting hypothesis is that the technique of hysteroscopy by vaporization would reduce the operative time by 30%. The number of subjects required per group will be 27 patients, or 54 patients in total over 24 months.

The expected results are a significant decrease in operative time with the vaporization hysteroscopy technique. This would be important because the reduction in operative time is associated with a reduction in complications of operative hysteroscopy and the possibility of treating larger fibroids with this technique.

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 18 years old.
* Non-pregnant patient
* A patient who had an ultrasound confirming the presence of a uterine fibroid to be treated less than 6 cm.
* Patient who had a diagnostic hysteroscopy confirming the presence of a uterine fibroid to be treated of type 0, 1 or 2 according to the FIGO classification.
* Patient presenting an indication for intra uterine fibroid resection (bleeding, fertility problems) by operative hysteroscopy.
* Patient having agreed to participate in the study and having signed an informed consent.

Exclusion Criteria:

* Minor patient
* Patient not affiliated to a social security system
* Persons benefiting from special protection: by virtue of articles L1121-5 to L1121-8 of the Public Health Code: pregnant or breast-feeding women, minors, adults under guardianship or curatorship, persons deprived of liberty.
* Patient refusing to sign the consent or unable to receive the information necessary to give informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 54 (Estimated)
Dates: Start 2021-09-25 (Actual); Primary Completion 2023-11-17 (Estimated); Study Completion 2024-05-17 (Estimated)

PRIMARY OUTCOMES:
Operative time | Baseline
  Operative time expressed in minutes

SECONDARY OUTCOMES:
The amount of distention fluid used during operative hysteroscopy | Baseline
  Measured by collection of the distention fluid pockets at the end of the procedure
Resection time | Baseline
  Time estimated in cm3/min based on ultrasound measurement of the volume of the myoma involved in the resection preoperatively and postoperatively, related to the operative time
Complication rate during operative hysteroscopy | Baseline
  Cervical tear rate and Rate of uterine perforations
The rate of discontinuation of the operative hysteroscopy before complete resection | Baseline
  Rate of discontinuation because of uterine perforations, operative time greater than 60 minutes, quantity of distension fluid greater than 9 liters, deficit of distension fluid greater than 1 liter, per operative haemorrhage
The rate of postoperative synechiae in patients of childbearing age. | between 6 and 8 weeks after the operation
  Rate of postoperative synechiae diagnosed at follow-up hysteroscopy in patients of childbearing age.
Operative pain | Baseline
  Operative pain evaluated by a visual analog scale (0-100mm). If the patient has a score of 0, it means that he/she has no pain. The higher the value, the more intense the pain.

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Director, Study Director — AP-HM
Locations (1):
- Assistance Publique Hôpitaux Marseille, Marseille, Bouches-du-Rhone, France

IPD SHARING:
Plan to Share IPD: No